CLINICAL TRIAL: NCT02016846
Title: Liraglutide Efficacy on Glucocorticoid Induced Hyperglycemia in Patients High Risk for Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Amit Tirosh, Dr, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0209-13
Record Dates: First submitted 2013-12-15; First posted 2013-12-20 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Glucocorticoid Induced Hyperglycemia
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Intervention (Active Comparator): Liraglutide, tapered from 0.6 mg/day to 1.8 mg/day.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide
  Arms: Intervention
Drug: Placebo
  Arms: Placebo

SUMMARY:
Glucocorticoids therapy exposes the patient to an increased risk for diabetes morbidity. However, there is no proven preventive therapy. GLP-1-RA has shown to improve glucose metabolism in healthy volunteers treated with glucocorticoids. We assume that GLP-1-RA will improve glucose metabolism in patients with high risk for diabetes morbidity, treated with glucocorticoids.

ELIGIBILITY:
Inclusion criteria:

* Planned treatment with T. Prednisone in dosage >0.5 mg/kg for two weeks or more.
* Age >18 years
* Body mass index >27 kg/m2 OR 1st degree relative with type 2 diabetes mellitus OR hypertension OR hyperlipidemia OR gestational diabetes in the past OR diagnosis of polycystic ovary syndrome.

Exclusion criteria:

* Glycosylated hemoglobin A1c >6.5%
* Diagnosis of diabetes mellitus or treatment with anti-glycemic drug
* Pancreatitis (acute or chronic) in the past
* Active malignancy
* Medullary thyroid carcinoma or multiple endocrine neoplasm type 2 of the patient or of 1st degree relative
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Glucose levels 2 hours after 75 gr OGTT | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Beilinson Campus, Petah Tikva, Israel